CLINICAL TRIAL: NCT01314872
Title: A Phase IIb Randomized, Placebo- and Active Comparator (Tolterodine)-Controlled, 2-Part Clinical Study of the Efficacy and Safety of MK-4618 in Patients With Overactive Bladder A 52-week Extension to: A Phase IIb Randomized, Placebo- and Active Comparator (Tolterodine)-Controlled, 2-Part Clinical Study of the Efficacy and Safety of MK-4618 in Patients With Overactive Bladder
Brief Title: A Study of the Efficacy and Safety of Vibegron (MK-4618) in Participants With Overactive Bladder (OAB) (MK-4618-008)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4618-008; 132241 (Registry Identifier: JAPIC-CTI); 2010-022121-15 (EudraCT Number); 2011-002533-18 (EudraCT Number)
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder; MK-4618; tolterodine
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (15):
- Part 1: placebo (Placebo Comparator): Participants received two placebo matching vibegron tablets and one placebo matching tolterodine extended release (ER) capsule, taken orally each morning, for 8 weeks.
  Interventions: Drug: Placebo matching vibegron; Drug: Placebo matching tolterodine ER
- Part 1: vibegron 3 mg (Experimental): Participants received one vibegron 3 mg tablet, one placebo matching vibegron tablet, and one placebo matching tolterodine ER capsule, taken orally each morning, for 8 weeks.
  Interventions: Drug: Vibegron; Drug: Placebo matching vibegron; Drug: Placebo matching tolterodine ER
- Part 1: vibegron 15 mg (Experimental): Participants received one vibegron 15 mg tablet, one placebo matching vibegron tablet, and one placebo matching tolterodine ER capsule, taken orally each morning, for 8 weeks.
  Interventions: Drug: Vibegron; Drug: Placebo matching vibegron; Drug: Placebo matching tolterodine ER
- Part 1: vibegron 50 mg (Experimental): Participants received one vibegron 50 mg tablet, one placebo matching vibegron tablet, and one placebo matching tolterodine ER capsule, taken orally each morning, for 8 weeks.
  Interventions: Drug: Vibegron; Drug: Placebo matching vibegron; Drug: Placebo matching tolterodine ER
- Part 1: vibegron 100 mg (Experimental): Participants received two vibegron 50 mg tablets and one placebo matching tolterodine ER capsule, taken orally each morning, for 8 weeks.
  Interventions: Drug: Vibegron; Drug: Placebo matching tolterodine ER
- Part 1: tolterodine ER 4 mg (Active Comparator): Participants received one tolterodine ER 4 mg capsule and two placebo matching vibegron tablets, taken orally each morning, for 8 weeks.
  Interventions: Drug: Tolterodine ER; Drug: Placebo matching vibegron
- Part 1: vibegron 50 mg + tolterodine ER 4 mg/vibegron 50 mg (Experimental): Participants received one vibegron 50 mg tablet and one placebo matching vibegron tablet, taken orally each morning, for 8 weeks. They also received one tolterodine ER 4 mg capsule for the first 4 weeks and one placebo matching tolterodine ER capsule for the second 4 weeks, both taken orally each morning.
  Interventions: Drug: Vibegron; Drug: Tolterodine ER; Drug: Placebo matching tolterodine ER
- Part 2: placebo (Placebo Comparator): Participants received two placebo matching vibegron tablets and one placebo matching tolterodine ER capsule, taken orally each morning, for 4 weeks.
  Interventions: Drug: Placebo matching vibegron; Drug: Placebo matching tolterodine ER
- Part 2: vibegron 100 mg (Experimental): Participants received two vibegron 50 mg tablets and one placebo matching tolterodine ER capsule, taken orally each morning, for 4 weeks.
  Interventions: Drug: Vibegron; Drug: Placebo matching tolterodine ER
- Part 2: tolterodine ER 4 mg (Active Comparator): Participants received one tolterodine ER 4 mg capsule and two placebo matching vibegron tablets, taken orally each morning, for 4 weeks.
  Interventions: Drug: Tolterodine ER; Drug: Placebo matching vibegron
- Part 2: vibegron 100 mg + tolterodine ER 4 mg (Experimental): Participants received two vibegron 50 mg tablets and one tolterodine ER 4 mg capsule, taken orally each morning, for 4 weeks.
  Interventions: Drug: Vibegron; Drug: Tolterodine ER
- Extension Study: vibegron 50 mg (Experimental): Participants in Base Study/Part 1 who received vibegron 50 mg continued their treatment in the Extension Study. In addition, participants in Base Study/Part 1 who received vibegron 3 mg received vibegron 50 mg in the Extension Study. Also, participants in Base Study/Part 1 who received vibegron 50 mg + tolterodine ER for 4 weeks, followed by vibegron 50 mg alone for 4 weeks, remained on vibegron 50 mg in the Extension Study. In the extension, participants received one vibegron 50 mg tablet, one placebo matching vibegron tablet, and one placebo matching tolterodine ER capsule, taken orally each morning, for 52 weeks.
  Interventions: Drug: Vibegron; Drug: Placebo matching vibegron; Drug: Placebo matching tolterodine ER
- Extension Study: vibegron 100 mg (Experimental): Participants in Base Study/Part 1 or Part 2 who received vibegron 100 mg continued their treatment in the Extension Study. In addition, participants in Base Study/Part 1 who received vibegron 15 mg received vibegron 100 mg in the Extension Study. In the extension, participants received two vibegron 50 mg tablets and one placebo matching tolterodine ER capsule, taken orally each morning, for 52 weeks.
  Interventions: Drug: Vibegron; Drug: Placebo matching tolterodine ER
- Extension Study: tolterodine ER 4 mg (Experimental): Participants in Base Study/Part 1 or Part 2 who received tolterodine ER 4 mg continued their treatment in the Extension Study. In addition, participants in Base Study/Part 1 who received placebo also received tolterodine ER 4 mg in the Extension Study. In the extension, participants received one tolterodine ER 4 mg capsule and two placebo matching vibegron tablets, taken orally each morning, for 52 weeks.
  Interventions: Drug: Tolterodine ER; Drug: Placebo matching vibegron
- Extension Study: vibegron 100 mg + tolterodine ER 4 mg (Experimental): Participants in Base Study/Part 1 who received vibegron 100 mg + tolterodine ER 4 mg continued their treatment in the Extension Study. In addition, participants in Base Study/Part 2 who received placebo were assigned to the vibegron 100 mg + tolterodine ER 4 mg arm in the Extension Study. In the extension, participants received two vibegron 50 mg tablets and one tolterodine ER 4 mg capsule, taken orally each morning, for 52 weeks.
  Interventions: Drug: Vibegron; Drug: Tolterodine ER

INTERVENTIONS:
Drug: Vibegron — Participants received vibegron oral tablets at dosages of 3 mg, 15 mg, 50 mg, or 100 mg depending on their vibegron arm assignment, taken orally each morning.
  Other Names: MK-4618
  Arms: Extension Study: vibegron 100 mg; Extension Study: vibegron 100 mg + tolterodine ER 4 mg; Extension Study: vibegron 50 mg; Part 1: vibegron 100 mg; Part 1: vibegron 15 mg; Part 1: vibegron 3 mg; Part 1: vibegron 50 mg; Part 1: vibegron 50 mg + tolterodine ER 4 mg/vibegron 50 mg; Part 2: vibegron 100 mg; Part 2: vibegron 100 mg + tolterodine ER 4 mg
Drug: Tolterodine ER — Participants received one tolterodine ER 4 mg capsule, taken orally once a day.
  Other Names: Detrol®
  Arms: Extension Study: tolterodine ER 4 mg; Extension Study: vibegron 100 mg + tolterodine ER 4 mg; Part 1: tolterodine ER 4 mg; Part 1: vibegron 50 mg + tolterodine ER 4 mg/vibegron 50 mg; Part 2: tolterodine ER 4 mg; Part 2: vibegron 100 mg + tolterodine ER 4 mg
Drug: Placebo matching vibegron — Participants received placebo matching vibegron tablets, taken orally each morning.
  Arms: Extension Study: tolterodine ER 4 mg; Extension Study: vibegron 50 mg; Part 1: placebo; Part 1: tolterodine ER 4 mg; Part 1: vibegron 15 mg; Part 1: vibegron 3 mg; Part 1: vibegron 50 mg; Part 2: placebo; Part 2: tolterodine ER 4 mg
Drug: Placebo matching tolterodine ER — Participants received placebo matching tolterodine ER capsule, taken orally each morning.
  Arms: Extension Study: vibegron 100 mg; Extension Study: vibegron 50 mg; Part 1: placebo; Part 1: vibegron 100 mg; Part 1: vibegron 15 mg; Part 1: vibegron 3 mg; Part 1: vibegron 50 mg; Part 1: vibegron 50 mg + tolterodine ER 4 mg/vibegron 50 mg; Part 2: placebo; Part 2: vibegron 100 mg

SUMMARY:
This is a 2-part study to assess if vibegron (MK-4618) reduces the number of daily urinations more effectively than placebo in participants with overactive bladder (OAB). The primary hypothesis of the base study is that administration of vibegron demonstrates a dose-related reduction, compared with placebo, in average number of daily micturitions in participants with OAB after 8 weeks of treatment.

DETAILED DESCRIPTION:
All participants received placebo (run-in) for 1 week prior to randomization to Parts 1 and 2. Participants who complete the base study may be screened for a year-long, multicenter extension for assessment of long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* If participant is of reproductive potential, must agree to remain abstinent or use (or have his/her partner use) 2 acceptable methods of birth control within the projected duration of the study
* Clinical history of OAB for at least 3 months and meets either the OAB wet or OAB dry criteria
* Is able to read, understand and complete questionnaires and voiding diaries without assistance
* Is ambulatory and in good general physical and mental health
* No clinically significant electrocardiogram or laboratory abnormality

Exclusion Criteria:

* If female, is currently pregnant or breast-feeding, or expecting to conceive within the projected duration of the study
* Evidence of diabetes insipidus, uncontrolled hyperglycemia or uncontrolled hypercalcemia
* Allergy, intolerance, or history of a significant clinical or laboratory adverse experience associated with any of the active or inactive components of tolterodine ER or vibegron (MK-4618) formulation; or has a history or active diagnosis of any condition contraindicated in the tolterodine ER prescribing label
* Has lower urinary tract pathology that could be responsible for urgency, frequency, or incontinence
* History of injury, surgery, or neurodegenerative diseases (e.g., multiple sclerosis) that could affect the lower urinary tract or its nerve supply
* History of continual urine leakage
* Surgery to correct stress urinary incontinence or pelvic organ prolapse within 6 months
* Known history of elevated postvoid residual
* Bladder training or electrostimulation within 2 weeks or is planning to initiate either procedure during the study
* Active or recurrent (>6 episodes per year) urinary tract infections
* Current hematuria
* Required use of an indwelling catheter or requires intermittent catheterization
* History of fecal incontinence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1395 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2012-10-22 (Actual); Study Completion 2013-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mitcheson HD, Samanta S, Muldowney K, Pinto CA, Rocha BA, Green S, Bennett N, Mudd PN Jr, Frenkl TL. Vibegron (RVT-901/MK-4618/KRP-114V) Administered Once Daily as Monotherapy or Concomitantly with Tolterodine in Patients with an Overactive Bladder: A Multicenter, Phase IIb, Randomized, Double-blind, Controlled Trial. Eur Urol. 2019 Feb;75(2):274-282. doi: 10.1016/j.eururo.2018.10.006. Epub 2018 Oct 25. PMID 30661513

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-Part, randomized, double blind placebo- and active-controlled, parallel-group study of vibegron in men and women with Overactive Bladder (OAB). Participants who enrolled in Part 1 were not eligible to participate in Part 2. Participants who completed Part 1 or Part 2 were eligible to enroll in an optional 1-year safety extension.
Period: Treatment Period 1
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg | Part 2: Placebo | Part 2: Vibegron 100 mg | Part 2: Tolterodine ER 4 mg | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Started | 141 | 144 | 134 | 150 | 149 | 135 | 134 | 64 | 112 | 122 | 110 | 0 | 0 | 0 | 0
Completed | 131 | 138 | 128 | 143 | 142 | 128 | 126 | 57 | 106 | 118 | 107 | 0 | 0 | 0 | 0
Not Completed | 10 | 6 | 6 | 7 | 7 | 7 | 8 | 7 | 6 | 4 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event, non-fatal | 4 | 2 | 3 | 2 | 2 | 4 | 4 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 2 | 3 | 1 | 3 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg | Part 2: Placebo | Part 2: Vibegron 100 mg | Part 2: Tolterodine ER 4 mg | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 223 | 248 | 240 | 134
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 175 | 188 | 187 | 110
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 48 | 60 | 53 | 24
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 12 | 9 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0
Not completed — Adverse event, non-fatal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 24 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 17 | 12 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg | Part 2: Placebo | Part 2: Vibegron 100 mg | Part 2: Tolterodine ER 4 mg | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg | Total
Number analyzed (Participants) | 141 | 144 | 134 | 150 | 149 | 135 | 134 | 64 | 112 | 122 | 110 | 1395
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (9.0) | 59.4 (8.7) | 58.6 (8.1) | 60.3 (8.7) | 60.3 (8.3) | 59.1 (8.1) | 59.4 (8.5) | 56.3 (10.6) | 57.2 (10.1) | 57.9 (10.9) | 55.5 (11.7) | 58.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 131 | 125 | 129 | 135 | 121 | 119 | 57 | 101 | 110 | 95 | 1251
  Male | 13 | 13 | 9 | 21 | 14 | 14 | 15 | 7 | 11 | 12 | 15 | 144

OUTCOME MEASURES:

1. Primary Outcome: Base Study/Part 1: Change From Baseline in Average Daily Micturitions at Week 8
Description: Participants were required to keep a voiding diary, recording the occurrence of each micturition. The average daily number of micturitions was calculated as the total number of micturitions that occurred over a week (4 to 10 days) during the Base Study, divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the average daily number of daily micturitions that occurred during the week of placebo run-in prior to Week 0 visit.
Time Frame: Baseline and Week 8
Population: Full analysis set population included all randomized participants who received at least one dose of study treatment and have either baseline data or at least one post-randomization observation for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Micturitions
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg
Number analyzed (Participants) | 141 | 144 | 132 | 148 | 148 | 134 | 134
Micturitions | -1.16 [-1.5 to -0.82] | -1.62 [-1.95 to -1.29] | -1.61 [-1.96 to -1.27] | -1.80 [-2.13 to -1.47] | -2.07 [-2.40 to -1.74] | -1.71 [-2.05 to -1.36] | -2.05 [-2.40 to -1.70]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: Vibegron 3 mg; Test type: Superiority or Other; p = 0.056, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, part and interaction of time by treatment; Difference in least squares (LS) means = -0.46, 95% CI 2-sided [-0.92 to 0.01]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: Vibegron 15 mg; Test type: Superiority or Other; p = 0.064, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, part and interaction of time by treatment; Difference in LS means = -0.45, 95% CI 2-sided [-0.93 to 0.03]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: Vibegron 50 mg; Test type: Superiority or Other; p = 0.007, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, part and interaction of time by treatment; Difference in LS means = -0.64, 95% CI 2-sided [-1.11 to -0.18]
Statistical Analysis 4: Comparison: Part 1: Placebo vs Part 1: Vibegron 100 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, part and interaction of time by treatment; Difference in LS means = -0.91, 95% CI 2-sided [-1.37 to -0.44]
Statistical Analysis 5: Comparison: Part 1: Placebo vs Part 1: Tolterodine ER 4 mg; Test type: Superiority or Other; p = 0.026, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, part and interaction of time by treatment; Difference in LS means = -0.54, 95% CI 2-sided [-1.02 to -0.07]

2. Primary Outcome: Base Study/Part 1 + Part 2: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug.
Time Frame: Part 1: up to 8 weeks; Part 2: up to 4 weeks. The time frame was an additional 2 weeks for participants not continuing to the Extension Study.
Population: All participants as treated population consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg | Part 2: Placebo | Part 2: Vibegron 100 mg | Part 2: Tolterodine ER 4 mg | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 141 | 144 | 134 | 148 | 149 | 135 | 134 | 64 | 112 | 122 | 110
Participants | 66 | 55 | 70 | 62 | 70 | 68 | 69 | 22 | 37 | 48 | 40

3. Primary Outcome: Base Study/Part 1 + Part 2: Number of Participants Who Had Study Medication Withdrawn Due to an AE
Description: as for outcome 2
Time Frame: Part 1: up to 8 weeks; Part 2: up to 4 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg | Part 2: Placebo | Part 2: Vibegron 100 mg | Part 2: Tolterodine ER 4 mg | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 141 | 144 | 134 | 148 | 149 | 135 | 134 | 64 | 112 | 122 | 110
Participants | 3 | 3 | 4 | 2 | 2 | 4 | 3 | 2 | 4 | 0 | 2

4. Primary Outcome: Extension Study: Number of Participants Who Experienced an Adverse Event (AE)
Description: as for outcome 2
Time Frame: Extension: up to 54 weeks (including 2-week follow-up)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 223 | 248 | 240 | 134
Participants | 134 | 157 | 158 | 82

5. Primary Outcome: Extension Study: Number of Participants Who Had Study Medication Withdrawn Due to an AE
Description: as for outcome 2
Time Frame: Extension: up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 223 | 248 | 240 | 134
Participants | 11 | 14 | 24 | 7

6. Secondary Outcome: Base Study/Part 1: Change From Baseline in Number of Urge Incontinence Episodes at Week 8
Description: Participants were required to keep a voiding diary, recording the occurrence of each total incontinence episode. The average daily number of total incontinence episodes was calculated as the total number of times a participant experienced such an episode over a week (4 to 10 days) during the Base Study, divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the average daily number of total incontinence episodes that occurred during the week of placebo run-in prior to Week 0 visit.
Time Frame: Baseline and Week 8
Population: Full analysis set population included all randomized participants who received at least one dose of study treatment and have either baseline data or at least one post-randomization observation for the analysis endpoint. This outcome measure included OAB Wet participants only.
Measure: Least Squares Mean (95% Confidence Interval); unit: Urge incontinence episodes
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg
Number analyzed (Participants) | 118 | 113 | 111 | 121 | 122 | 100 | 111
Urge incontinence episodes | -1.24 [-1.52 to -0.95] | -1.52 [-1.81 to -1.23] | -1.81 [-2.10 to -1.51] | -1.95 [-2.23 to -1.67] | -1.95 [-2.23 to -1.67] | -1.69 [-2.00 to -1.38] | -1.71 [-2.01 to -1.42]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: Vibegron 3 mg; Test type: Superiority or Other; p = 0.167, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.28, 95% CI 2-sided [-0.68 to 0.12]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: Vibegron 15 mg; Test type: Superiority or Other; p = 0.005, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.57, 95% CI 2-sided [-0.97 to -0.17]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: Vibegron 50 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.72, 95% CI 2-sided [-1.11 to -0.33]
Statistical Analysis 4: Comparison: Part 1: Placebo vs Part 1: Vibegron 100 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.71, 95% CI 2-sided [-1.10 to -0.32]
Statistical Analysis 5: Comparison: Part 1: Placebo vs Part 1: Tolterodine ER 4 mg; Test type: Superiority or Other; p = 0.030, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.46, 95% CI 2-sided [-0.87 to -0.04]

7. Secondary Outcome: Base Study/Part 1: Change From Baseline in Average Daily Number of Total Incontinence Episodes at Week 8
Description: as for outcome 6
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Incontinence episodes
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg
Number analyzed (Participants) | 118 | 113 | 111 | 121 | 122 | 100 | 111
Incontinence episodes | -1.52 [-1.84 to -1.21] | -1.71 [-2.02 to -1.39] | -2.01 [-2.33 to -1.69] | -2.13 [-2.43 to -1.82] | -2.11 [-2.41 to -1.80] | -1.86 [-2.20 to -1.52] | -2.00 [-2.32 to -1.68]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: Vibegron 3 mg; Test type: Superiority or Other; p = 0.401, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS Means = -0.18, 95% CI 2-sided [-0.61 to 0.25]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: Vibegron 15 mg; Test type: Superiority or Other; p = 0.029, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS Means = -0.48, 95% CI 2-sided [-0.91 to -0.05]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: Vibegron 50 mg; Test type: Superiority or Other; p = 0.005, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS Means = -0.60, 95% CI 2-sided [-1.02 to -0.18]
Statistical Analysis 4: Comparison: Part 1: Placebo vs Part 1: Vibegron 100 mg; Test type: Superiority or Other; p = 0.007, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS Means = -0.58, 95% CI 2-sided [-1.01 to -0.16]
Statistical Analysis 5: Comparison: Part 1: Placebo vs Part 1: Tolterodine ER 4 mg; Test type: Superiority or Other; p = 0.140, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS Means = -0.34, 95% CI 2-sided [-0.78 to 0.11]

8. Secondary Outcome: Base Study/Part 1: Change From Baseline in Average Daily Number of Strong Urge Episodes at Week 8
Description: Participants were required to keep a voiding diary, recording the occurrence of each strong urge episode. The average daily number of strong urge episodes was calculated as the total number of times a participant experienced such an episode over a week (4 to 10 days) during the Base Study, divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the average daily number of strong urge episodes that occurred during the week of placebo run-in prior to Week 0 visit.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Strong urge episodes
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg
Number analyzed (Participants) | 141 | 144 | 132 | 148 | 148 | 134 | 134
Strong urge episodes | -1.59 [-2.07 to -1.11] | -1.77 [-2.24 to -1.30] | -2.27 [-2.76 to -1.78] | -2.36 [-2.82 to -1.89] | -2.83 [-3.30 to -2.37] | -2.53 [-3.03 to -2.04] | -2.73 [-3.22 to -2.24]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: Vibegron 3 mg; Test type: Superiority or Other; p = 0.598, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.18, 95% CI 2-sided [-0.84 to 0.49]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: Vibegron 15 mg; Test type: Superiority or Other; p = 0.052, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.67, 95% CI 2-sided [-1.35 to 0.01]
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: Vibegron 50 mg; Test type: Superiority or Other; p = 0.024, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.76, 95% CI 2-sided [-1.43 to -0.10]
Statistical Analysis 4: Comparison: Part 1: Placebo vs Part 1: Vibegron 100 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -1.24, 95% CI 2-sided [-1.90 to -0.58]
Statistical Analysis 5: Comparison: Part 1: Placebo vs Part 1: Tolterodine ER 4 mg; Test type: Superiority or Other; p = 0.007, Constrained Longitudinal Data Analysis; Constrained longitudinal data analysis model includes terms for time, region, and interaction of time by treatment; Difference in LS means = -0.94, 95% CI 2-sided [-1.62 to -0.26]

9. Secondary Outcome: Extension Study: Change From Baseline in Average Daily Micturitions at Week 52
Description: Participants were required to keep a voiding diary, recording the daily occurrence of each micturition. The average daily number of micturitions was calculated as the total number of recorded micturitions that occurred during the 52-week Extension Study, divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the value at Week 0 of the Base Study.
Time Frame: Baseline and Week 52 of Extension Study
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Micturitions
Arm/Group | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 223 | 246 | 240 | 134
Micturitions | -2.53 [-2.87 to -2.20] | -2.77 [-3.08 to -2.45] | -2.15 [-2.47 to -1.83] | -3.25 [-3.67 to -2.83]
Statistical Analysis 1: Comparison: Extension Study: Vibegron 100 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = -0.49, 95% CI 2-sided [-1.00 to 0.03]
Statistical Analysis 2: Comparison: Extension Study: Tolterodine ER 4 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = -1.10, 95% CI 2-sided [-1.62 to -0.58]

10. Secondary Outcome: Extension Study: Change From Baseline in Average Daily Number of Urge Incontinence Episodes at Week 52
Description: Participants were required to keep a voiding diary, recording the occurrence of each urge incontinence episode. The average daily number of urge incontinence episodes was calculated as the total number of times a participant experienced such an episode during 52-week Extension Study, divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the value at Week 0 of the Base Study.
Time Frame: Baseline and Week 52 of Extension Study
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Urge incontinence episodes
Arm/Group | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 179 | 200 | 189 | 112
Urge incontinence episodes | -2.43 [-2.72 to -2.14] | -2.15 [-2.43 to -1.87] | -2.23 [-2.51 to -1.94] | -2.44 [-2.79 to -2.09]
Statistical Analysis 1: Comparison: Extension Study: Vibegron 100 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = -0.29, 95% CI 2-sided [-0.71 to 0.13]
Statistical Analysis 2: Comparison: Extension Study: Tolterodine ER 4 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = -0.21, 95% CI 2-sided [-0.64 to 0.21]

11. Secondary Outcome: Extension Study: Change From Baseline in Average Daily Number of Total Incontinence Episodes at Week 52
Description: Participants were required to keep a voiding diary, recording the occurrence of each total incontinence episode. The average daily number of total incontinence episodes was calculated as the total number of times a participant experienced such an episode during 52-week Extension Study, divided by the total divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the value at Week 0 of the Base Study.
Time Frame: Baseline and Week 52 of Extension Study
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Incontinence episodes
Arm/Group | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 179 | 200 | 189 | 112
Incontinence episodes | -2.70 [-3.03 to -2.36] | -2.42 [-2.74 to -2.09] | -2.50 [-2.83 to -2.17] | -2.48 [-2.89 to -2.07]
Statistical Analysis 1: Comparison: Extension Study: Vibegron 100 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = -0.07, 95% CI 2-sided [-0.56 to 0.43]
Statistical Analysis 2: Comparison: Extension Study: Tolterodine ER 4 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = 0.02, 95% CI 2-sided [-0.48 to 0.51]

12. Secondary Outcome: Extension Study: Change From Baseline in Average Daily Number of Strong Urge Episodes at Week 52
Description: Participants were required to keep a voiding diary, recording the occurrence of each strong urge episode. The average daily number of strong urge episodes was calculated as the total number of times a participant experienced such an episode during 52-week Extension Study, divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the value at Week 0 of the Base Study.
Time Frame: Baseline and Week 52 of Extension Study
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Strong urge episodes
Arm/Group | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg
Number analyzed (Participants) | 223 | 246 | 240 | 134
Strong urge episodes | -3.11 [-3.55 to -2.67] | -3.42 [-3.84 to -3.00] | -2.94 [-3.36 to -2.52] | -4.18 [-4.74 to -3.63]
Statistical Analysis 1: Comparison: Extension Study: Vibegron 100 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = -0.76, 95% CI 2-sided [-1.45 to -0.08]
Statistical Analysis 2: Comparison: Extension Study: Tolterodine ER 4 mg vs Extension Study: Vibegron 100 mg + Tolterodine ER 4 mg; Test type: Superiority or Other; Difference in LS means = -1.24, 95% CI 2-sided [-1.93 to -0.56]

ADVERSE EVENTS:
Time Frame: Part 1: up to approximately 10 weeks (including 2 week follow-up unless entering extension); Part 2: up to approximately 6 weeks (including 2 week follow-up unless entering extension); Extension: up to approximately 54 weeks (including 2 week follow-up)
Description: All participants as treated population consists of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received. Two participants who were randomized but not treated were excluded from the Part 1: vibegron 50 mg arm.
Groups:
- Extension Study: Vibegron 50 mg + Tolterodine ER 4 mg: Participants in Base Study/Part 1 who received vibegron 100 mg + tolterodine ER 4 mg continued their treatment in the Extension Study. In addition, participants in Base Study/Part 2 who received placebo were assigned to the vibegron 100 mg + tolterodine ER 4 mg arm in the Extension Study. In the extension, participants received two vibegron 50 mg tablets and one tolterodine ER 4 mg capsule, taken orally each morning, for 52 weeks.
Arm/Group | Part 1: Placebo | Part 1: Vibegron 3 mg | Part 1: Vibegron 15 mg | Part 1: Vibegron 50 mg | Part 1: Vibegron 100 mg | Part 1: Tolterodine ER 4 mg | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg | Part 2: Placebo | Part 2: Vibegron 100 mg | Part 2: Tolterodine ER 4 mg | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg | Extension Study: Vibegron 50 mg | Extension Study: Vibegron 100 mg | Extension Study: Tolterodine ER 4 mg | Extension Study: Vibegron 50 mg + Tolterodine ER 4 mg
Serious Adverse Events (participants affected / at risk) | 2/141 | 1/144 | 0/134 | 1/148 | 0/149 | 1/135 | 1/134 | 0/64 | 0/112 | 2/122 | 0/110 | 14/223 | 8/248 | 18/240 | 1/134
Other Adverse Events (participants affected / at risk) | 32/141 | 21/144 | 27/134 | 30/148 | 33/149 | 33/135 | 27/134 | 6/64 | 5/112 | 21/122 | 20/110 | 59/223 | 73/248 | 70/240 | 38/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=141) | Part 1: Vibegron 3 mg (N=144) | Part 1: Vibegron 15 mg (N=134) | Part 1: Vibegron 50 mg (N=148) | Part 1: Vibegron 100 mg (N=149) | Part 1: Tolterodine ER 4 mg (N=135) | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg (N=134) | Part 2: Placebo (N=64) | Part 2: Vibegron 100 mg (N=112) | Part 2: Tolterodine ER 4 mg (N=122) | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg (N=110) | Extension Study: Vibegron 50 mg (N=223) | Extension Study: Vibegron 100 mg (N=248) | Extension Study: Tolterodine ER 4 mg (N=240) | Extension Study: Vibegron 50 mg + Tolterodine ER 4 mg (N=134)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gatrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Devise dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Periarthirits (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascluar accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Loss of conciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=141) | Part 1: Vibegron 3 mg (N=144) | Part 1: Vibegron 15 mg (N=134) | Part 1: Vibegron 50 mg (N=148) | Part 1: Vibegron 100 mg (N=149) | Part 1: Tolterodine ER 4 mg (N=135) | Part 1: Vibegron 50 mg + Tolterodine ER 4 mg/Vibegron 50 mg (N=134) | Part 2: Placebo (N=64) | Part 2: Vibegron 100 mg (N=112) | Part 2: Tolterodine ER 4 mg (N=122) | Part 2: Vibegron 100 mg + Tolterodine ER 4 mg (N=110) | Extension Study: Vibegron 50 mg (N=223) | Extension Study: Vibegron 100 mg (N=248) | Extension Study: Tolterodine ER 4 mg (N=240) | Extension Study: Vibegron 50 mg + Tolterodine ER 4 mg (N=134)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 4 (4) | 2 (2) | 1 (1) | 5 (5) | 7 (8) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 9 (9) | 9 (10) | 10 (10) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 5 (5) | 6 (6) | 7 (8) | 3 (3) | 14 (14) | 11 (11) | 4 (4) | 1 (1) | 8 (8) | 13 (14) | 8 (8) | 8 (8) | 18 (18) | 6 (6)
Nasopharyngitis (Infections and infestations) | 14 (15) | 3 (3) | 7 (8) | 8 (9) | 6 (6) | 3 (3) | 3 (4) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 12 (18) | 24 (30) | 20 (25) | 15 (19)
Urinary tract infection (Infections and infestations) | 5 (5) | 5 (5) | 5 (5) | 8 (8) | 6 (6) | 4 (5) | 7 (8) | 2 (2) | 2 (2) | 8 (8) | 5 (5) | 27 (42) | 22 (33) | 27 (44) | 8 (8)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 6 (6) | 4 (5) | 11 (11) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (8) | 4 (4) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 3 (3) | 6 (6) | 6 (8) | 10 (13) | 4 (4) | 6 (7) | 2 (4) | 2 (2) | 5 (6) | 7 (7) | 13 (13) | 4 (4) | 6 (7) | 5 (5)
Constipation (Gastrointestinal disorders) | 3 (4) | 5 (5) | 6 (6) | 6 (6) | 1 (1) | 4 (4) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 7 (7) | 9 (9) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 9 (9) | 14 (14) | 10 (10) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.